## The University of Hong Kong Department of Social Work and Social Administration

# The Implementation of Cognitive Stimulation Therapy Hong Kong Version (CST-HK) for Promoting Cognitive Functioning and Psychosocial Well-being of People with Dementia

Joint Informed Consent for People with Dementia and their Caregiver

You are invited to participate in this research study conducted by Dr. Gloria Wong from Department of Social Work and Social Administration, The University of Hong Kong. Your participation in this study is entirely voluntary. You should read the information below, and ask questions about anything you do not understand, before deciding whether to participate.

#### Purpose of Study

The research aims to (1) investigate the effectiveness of CST-HK among people with mild-to-moderate cognitive impairment in Hong Kong in a larger scale across service settings and to (2) explore the effectiveness of CST-HK delivered by non-professional staff, as a possible solution to address the shortage of specialized healthcare manpower and increasing demands of non-pharmacological interventions for people with dementia.

#### **Procedures**

Cognitive stimulation therapy (CST) is an evidence-based intervention, which is recommended for people with Alzheimer Disease from early to moderate stages in the UK. CST-HK is the revised version with cultural adaptation for HK. It is a group-based intervention (45 mins per session, two times a week, for 7 weeks in total). You or your family member will receive the 14-session group CST-HK. Before and after attending the group CST-HK, it will take you and your family members 45 mins respectively undergoing a clinical interview and some assessments, including demographic information, cognitive functioning and other psychosocial assessments. In the process of the intervention, researchers will conduct the on-site observation. Your understanding and approval of the procedures of the study is required if you are to participate in this study.

#### **Potential Benefits**

You may receive no medical benefit from participating in this study directly. However, your participation will contribute towards our understanding and future development of non-pharmacological interventions in HK for people with dementia.

## **Privacy and Confidentiality**

Any record or information obtained in this study will be treated as strictly confidential, will be known to no one except members of the research team, and will be used for research purposes only. Each participant's identity will be kept in anonymity during the data record and analysis processes. To ensure anonymity, a specified code, containing no personal information, will be assigned as an identifier to each participant in the study. Participants will not be identified by name in any report of the completed study. The anonymized data obtained in this study will be retained for up to 5 years, and will be destroyed subsequently after.

#### Participation and Withdrawal

All participants in the captioned research project is on a voluntary basis, and retains the right to refuse participation or withdraw from the captioned research project at any time without any consequences or any loss of benefits that the participant is otherwise entitled to receive. When you participate in the study, the current care you or your family member are receiving will be provided as usual. During the intervention, you can stop participating at any time if you or your family discomfort. Considering the safety and wellbeing of participants, researchers may also terminate your or your family member's participation in the study. If the decision is made, you and your family member will be informed ahead.

## **Questions and Concerns**

You may withdraw your consent at any time and discontinue participation without penalty. You are not waiving any legal claims or rights because of your participation in this research study. If you have any further questions or enquiries, please do not hesitate to contact our research coordinator, Mr. Chung, Yui Ching (Tel: +852-2708-3677; Email: brianchung@ywca.org.hk). If you wish to know more about the rights as a research participant, please do not hesitate to contact the Human Research Ethics Committee for Non-Clinical Faculties (HREC), the University of Hong Kong (Tel: +852-2241-5267).

| Signature o | f Research | <b>Participants</b> |
|-------------|------------|---------------------|

| | | Please initial | box |
|---|---|---|---|
| have read, or someone has read to me, and I understand the information provided above. | | | |
| | to ask questions and all my que | estions have been answered to my | |
| satisfaction. | | | |
| | - | to withdraw at any time without | |
| negative consequences or benefits l | | | |
| I have been given a copy of this form | | | Ш |
| I willingly agree for my family me | ember and myself to participate | in the research it describes. | |
| | | ed by the HKU research team after nation about related studies in the | |
| Name of Participant | Signature of Participant | Date | |
| Name of Caregiver | Signature of Caregiver | Date | |
| Signature of Investigator | | | |
| I have explained the research to the | he subject and answered all his or | her questions. I believe that he or | |
| she understands the information of | · | • | |
| | | , | |
| Name of Investigator | Signature of Investigator | <br>Date | |